CLINICAL TRIAL: NCT07308392
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase II Clinical Trial Evaluating the Efficacy and Safety of HRS-7249 and SHR-1918 in Patients With Severe Hypertriglyceridemia at High Risk of Acute Pancreatitis.
Brief Title: Phase II Clinical Trial Evaluating the Efficacy and Safety of HRS-7249 and SHR-1918 in Patients With Severe Hypertriglyceridemia at High Risk of Acute Pancreatitis
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fujian Shengdi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HRS-7249-202
Record Dates: First submitted 2025-12-15; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-11

CONDITIONS: Severe Hypertriglyceridemia With a High Risk of Acute Pancreatitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HRS-7249 injection (Experimental)
  Interventions: Drug: HRS-7249 injection set
- HRS-7249 injection placebo (Placebo Comparator)
  Interventions: Drug: HRS-7249 injection placebo set
- SHR-1918 injection (Experimental)
  Interventions: Drug: SHR-1918 injection set
- SHR-1918 injection placebo (Placebo Comparator)
  Interventions: Drug: SHR-1918 injection placebo set

INTERVENTIONS:
Drug: HRS-7249 injection set — HRS-7249 injection set
  Arms: HRS-7249 injection
Drug: SHR-1918 injection set — SHR-1918 injection set
  Arms: SHR-1918 injection
Drug: HRS-7249 injection placebo set — HRS-7249 injection placebo set
  Arms: HRS-7249 injection placebo
Drug: SHR-1918 injection placebo set — SHR-1918 injection placebo set
  Arms: SHR-1918 injection placebo

SUMMARY:
Phase II clinical trial evaluating the efficacy and safety of HRS-7249 and SHR-1918 in patients with severe hypertriglyceridemia at high risk of acute pancreatitis

ELIGIBILITY:
Inclusion Criteria:

1. Understand the research procedures and methods, voluntarily participate in this trial, and sign the informed consent form in writing;
2. Male or female aged ≥18 years and <80 years on the day of signing the informed consent form.

Exclusion Criteria:

1. History of gallstones at the time of screening or previously (except for patients who had their gallbladder removed more than 3 months ago);
2. Acute pancreatitis that has clinically recovered ≤4 weeks before screening or randomization;
3. Malignant tumor within 5 years before screening or randomization (except for non-melanoma skin cancer or cervical carcinoma in situ that has been radically treated);
4. Grade 3/4 heart failure at the time of screening or before randomization;
5. Acute coronary syndrome (such as myocardial infarction, unstable angina), history of coronary artery bypass grafting, percutaneous coronary intervention, peripheral artery revascularization, cerebrovascular diseases (such as stroke, transient ischemic attack), heart failure hospitalization, etc., within 3 months before screening or randomization;
6. Severe arrhythmias within 3 months before screening or randomization, such as recurrent symptomatic frequent ventricular premature beats, ventricular tachycardia, atrial fibrillation with rapid ventricular rate;
7. Severe infection within 3 months before screening;
8. History or presence of nephrotic syndrome, severe liver disease, Cushing's syndrome, or other diseases significantly affecting lipid levels at screening;
9. History or presence of hyperthyroidism or hypothyroidism at screening;
10. Poorly controlled hypertension at screening or before randomization (systolic blood pressure ≥180 mmHg and/or diastolic blood pressure ≥110 mmHg);
11. Diabetes with any of the following: a. Newly diagnosed within 12 weeks before screening or randomization; b. HbA1c ≥8.0% at screening; c. Type 1 diabetes;
12. Unstable or severe liver, kidney, cardiovascular, psychiatric, neurological, endocrine, hematologic, or other diseases at screening or before randomization, where the investigator determines participation poses an unacceptable risk to the subject;
13. Serious trauma or major surgery within 6 months before screening, or planning major surgery during the trial;
14. Plasma exchange therapy within 4 weeks before screening or randomization, or planned during the trial;
15. Use of other drugs significantly affecting lipid levels within 4 weeks before screening or randomization, or planned during the trial, such as traditional Chinese medicine containing statins (e.g., Zhibituo, Zhibitai), other lipid-lowering drugs and supplements (e.g., probucol, bile acid sequestrants, niacin, over-the-counter drugs, red yeast rice), GLP-1 agonists, other incretin analogues;
16. Use of weight-loss drugs or undergoing weight-altering surgery within 2 months before screening or randomization, or planned during the study;
17. History of drug abuse or alcohol abuse (including heavy drinking [average ethanol intake >80 g/day], previously diagnosed alcohol harmful use, alcohol dependence, alcohol poisoning, alcohol withdrawal, alcohol-related disorder, or alcohol-induced psychiatric or behavioral disorder);
18. Significant lifestyle changes within 4 weeks before screening or randomization, or refusal to follow lifestyle guidance or limit alcohol intake to <30 g/day during the study;
19. eGFR calculated by the Modification of Diet in Renal Disease (MDRD) formula <60 mL/min/1.73 m²;
20. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥3 times the upper limit of normal (ULN);
21. Total bilirubin or direct bilirubin ≥2 times ULN;
22. Creatine kinase (CK) >1.5 times ULN;
23. Platelet count <100 x 10⁹/L (or history of thrombocytopenia);
24. Hemoglobin <60 g/L;
25. Confirmed active syphilis, positive test result for human immunodeficiency virus antibody (HIV-Ab) or hepatitis C virus antibody (HCV-Ab), positive hepatitis B surface antigen (HBsAg) with HBV-DNA ≥1000 copies/ml (or ≥200 IU/ml, or if the detection lower limit is higher than 1000 copies/ml or 200 IU/ml, HBV-DNA ≥ detection lower limit);
26. Thyroid-stimulating hormone (TSH) below the lower limit of normal (LLN) or above 1.5 times ULN;
27. Participation in any interventional drug clinical trial within 3 months prior to screening (participation is defined as administration of the investigational product to the subject), or still within 5 half-lives of the investigational product before screening, whichever is longer; previous participation in non-interventional clinical trials or device-related clinical trials may be judged by the investigator for inclusion;
28. Pregnant or breastfeeding women;
29. Women of childbearing potential who have not used contraception within 30 days prior to screening; women of childbearing potential and male subjects with partners of childbearing age who refuse to avoid donating sperm/eggs from the time of signing the informed consent until the end of the follow-up period, or refuse to comply with relevant contraceptive requirements;
30. Other conditions deemed by the investigator to make the subject unsuitable for participation in the trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Percentage change in mean TG from baseline at weeks 44 and 48 of treatment | at 44＆48 weeks after the start of administration
Proportion of subjects experiencing AP during the double-blind treatment period | within 48 weeks after the start of administration

SECONDARY OUTCOMES:
During the double-blind treatment period, the time and severity of the first occurrence of AP | within 48 weeks after the start of administration
During the double-blind treatment period, the proportion of subjects who developed HTG-AP, the time to first occurrence of HTG-AP, and its severity | within 48 weeks after the start of administration

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University (Jiangsu Provincial People's Hospital), Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided